CLINICAL TRIAL: NCT00075192
Title: A Phase 1, Open Label, Non-Randomized, Dose Escalation Study to Evaluate the Safety of CP-675,206 in Combination With Neoadjuvant Androgen Ablation and a Phase 2, Open Label, Randomized Study to Evaluate the Efficacy of CP-675,206 in Combination With Neoadjuvant Androgen Ablation and Androgen Ablation Alone in Patients With High Risk Prostate Cancer
Brief Title: CP-675,206 With Neoadjuvant Hormone Therapy in Patients With High Risk Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671004
Record Dates: First submitted 2004-01-05; First posted 2004-01-07 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tremelimumab; Leuprolide; bicalutamide

INTERVENTIONS:
Drug: CP-675,206 and leuprolide acetate and bicalutamide
Drug: leuprolide acetate and bicalutamide

SUMMARY:
This is a multi-center, open label, randomized study. Patients will be randomized to one of the following arms with an allocation ratio of 3:1, respectively: Arm A: CP-675,206 + neoadjuvant hormone therapy (NHT) OR Arm B: neoadjuvant hormone therapy. After randomization, patients will receive study treatment for three cycles (one cycle is defined as 28 days). After completion of three cycles, patients will undergo a prostatectomy and pathology assessments will be completed at a central laboratory, the Armed Forces Institute of Pathology (AFIP) in Washington, DC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, previously untreated
* Potential candidate for radical prostatectomy on the basis of the patient's general medical condition, performance status, and life expectancy
* Potential candidate for NHT prior to prostatectomy, including high or intermediate risk of recurrence, based on an estimated risk of biochemical recurrence: High risk category: PSA >20 or Gleason score 8 or cT2c/cT3 OR Intermediate risk category: PSA >10 and d20 or Gleason score 7 or cT2b
* No evidence of metastatic disease by physical examination, bone scan, and computed tomography, or MRI, of the abdomen and pelvis
* Age > 18 years
* ECOG performance status 0-1
* Adequate bone marrow, hepatic, and renal function determined within 2 weeks prior to starting therapy
* Availability of prostatectomy specimen for histological analysis at the Armed Forces Institute of Pathology

Exclusion Criteria:

* Prior hormone therapy, radiation, chemotherapy, or immunologic therapy for prostate cancer
* History of, or significant risk for, chronic inflammatory or autoimmune disease
* Potential requirement for systemic corticosteroids before surgery based on prior history
* History of autoimmune colitis or chronic GI conditions associated with diarrhea or bleeding, or current acute colitis of any origin
* Any serious uncontrolled medical disorder or active infection which would impair ability to receive study treatment and subsequent prostatectomy
* Coexisting malignancies except basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Assess safety of combination therapy and effectiveness as assessed by pathological response after 3 months of treatment follow for disease status for a maximum of 24 months

SECONDARY OUTCOMES:
assess Pk during treatment monitor for human anti-human antibodies at the end of the study explore genetic influences on safety and/or immune response

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, La Masa, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gallatin, Tennessee
  - Research Site, Hermitage, Tennessee
  - Research Site, Lebanon, Tennessee
  - Research Site, Murfreesboro, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Smyrna, Tennessee